CLINICAL TRIAL: NCT06817785
Title: Soft Lens Study: Biomedics 1 Day Extra Sphere and Clariti 1 Day Sphere
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision International Limited (CVIL) (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EX-MKTG-164
Record Dates: First submitted 2025-02-05; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens 1 (ocufilcon D) (Experimental): All participants will wear lens 1 for 15 minutes (Period 1).
  Interventions: Device: Lens 1 (ocufilcon D)
- Lens 2 (somofilcon A) (Experimental): All participants will wear lens 2 for 15 minutes (Period 2).
  Interventions: Device: Lens 2 (somofilcon A)

INTERVENTIONS:
Device: Lens 1 (ocufilcon D) — 15 minutes of daily wear
  Arms: Lens 1 (ocufilcon D)
Device: Lens 2 (somofilcon A) — 15 minutes of daily wear
  Arms: Lens 2 (somofilcon A)

SUMMARY:
The aim of this study is to evaluate and compare the performance of two soft contact lenses.

DETAILED DESCRIPTION:
The aim of this study is to evaluate and compare the performance of a hydrogel lens and a silicone hydrogel lens in existing myopic soft lens wearers.

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years of age and have full legal capacity to volunteer;
2. Have understood and signed an information consent letter;
3. Are willing and able to maintain the appointment schedule;
4. Are an adapted soft contact lens wearer;
5. Have a vertex-corrected contact lens prescription of -1.00DS to -6.00DS (inclusive) in each eye;
6. Have a refraction with a cylinder component of no more than -1.00DC in each eye;
7. Can be fitted with and achieve a distance visual acuity of +0.10 logMAR or better in each eye with the study contact lenses.

Exclusion Criteria:

1. Are participating in any concurrent clinical or research study;
2. Have any known active ocular disease and/or infection or slit lamp findings that would contraindicate contact lens use;
3. Have a systemic condition that would contraindicate contact lens use;
4. Are using any systemic or topical medications that would contraindicate contact lens use;
5. Have known sensitivity to the diagnostic fluorescein sodium to be used in the study;
6. Are an employee of the Centre for Ocular Research & Education directly involved in the study (i.e. on the delegation log).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2025-02-21 (Estimated); Study Completion 2025-02-21 (Estimated)

PRIMARY OUTCOMES:
Lens Comfort | Immediately after lens application
  The primary outcome of this study is lens comfort immediately after lens application on a scale of 0-100 (0= worst, 100=best).

CONTACTS AND LOCATIONS:
Overall Officials: Lyndon Jones, PhD FCOptom, Principal Investigator — Centre for Ocular Research and Education
Locations (1):
- School of Optometry and Vision Science, Waterloo, Ontario, Canada